CLINICAL TRIAL: NCT06070662
Title: Non-invasive Diagnosis of Coronary Microvascular Disease Using Novel CMR and CT Techniques: a Pilot Study
Brief Title: Non-invasive Diagnosis of Coronary Microvascular Disease: Pilot Study
Status: Recruiting | Type: Observational
Sponsor: University of Leicester (Other)
Responsible Party: Sponsor
Other Study IDs: 0844
Record Dates: First submitted 2022-03-25; First posted 2023-10-06 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Microvascular Angina
Keywords: Coronary microvascular disease; Angina; Non-invasive testing
MeSH Terms: conditions — Microvascular Angina; Angina Pectoris

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suspected coronary microvascular disease confirmed at angiography (expected n=8): Individuals with suspected coronary microvascular disease based on CT and MRI scans completed as part of the main research study. Those with confirmed coronary microvascular disease will complete an MRI scan as part of this pilot study and their CT scan will undergo additional analysis.
  Interventions: Diagnostic Test: Coronary microvascular disease testing during coronary angiography; Diagnostic Test: Cardiac magnetic resonance scan including exercise; Diagnostic Test: Additional analysis of already acquired CT scan
- Suspected coronary microvascular disease not confirmed at angiography (expected n=4): Individuals with suspected coronary microvascular disease based on CT and MRI scans completed as part of the main research study. If this is not confirmed coronary microvascular disease they will not undergo any further investigations as part of this research study.
  Interventions: Diagnostic Test: Coronary microvascular disease testing during coronary angiography
- Multivessel coronary artery disease (n=12): Individuals with multivessel coronary artery disease, diagnosed based on CT and MRI scans completed as part of the main research study and confirmed at angiography.
  Interventions: Diagnostic Test: Coronary microvascular disease testing during coronary angiography; Diagnostic Test: Cardiac magnetic resonance scan including exercise; Diagnostic Test: Additional analysis of already acquired CT scan

INTERVENTIONS:
Diagnostic Test: Coronary microvascular disease testing during coronary angiography — During invasive coronary angiography, in addition to coronary angiography performed as per routine clinical care, participants will have angiographic testing for coronary microvascular disease using routine clinical procedures. This will consist of fractional flow reserve (FFR), coronary flow reserve, index of microvascular resistance and vasospasm provocation testing with acetylcholine (Ach).
Diagnostic Test: Cardiac magnetic resonance scan including exercise — Participants will undergo a cardiac magnetic resonance scan compromising 1) T1 mapping, 2) oxygenation-sensitive MRI and 3) perfusion imaging. All will be obtained at rest and during exercise using a step ergometer.
  Groups: Multivessel coronary artery disease (n=12); Suspected coronary microvascular disease confirmed at angiography (expected n=8)
Diagnostic Test: Additional analysis of already acquired CT scan — Previously acquired CTCA images from the main research study will be transferred to Heartflow for computation of coronary blood volume.
  Groups: Multivessel coronary artery disease (n=12); Suspected coronary microvascular disease confirmed at angiography (expected n=8)

SUMMARY:
* 40% of patients presenting with stable chest pain (angina) have no significant blockage of the main heart arteries. Identifying why these patients have symptoms will mean better treatment options can be developed.
* About 60% of these patients have evidence of coronary microvascular disease (CMD). In this condition there is a problem with the heart's microvessels (very small blood vessels that branch from the main heart arteries). Due to problems with these vessels there is a mismatch between the blood supply to the heart and its oxygen consumption, causing chest pain and this can also lead to major heart events.
* At present, to diagnose this condition, specialised techniques during an invasive test, called a coronary angiogram, are required. As this is an invasive test, it can be lead to complications and cause discomfort.
* Non-invasive ways of diagnosing CMD are required to improve the diagnosis and management of this condition.
* This study aims to provide initial data on whether novel imaging techniques using CT and MRI scans, which are much less invasive, could identify CMD.
* To do this, patients with suspected angina referred for angiography and who are already participants in the main research study 'CMR versus CT-FFR in CAD' study will be recruited.
* These will be patients with suspected CMD and also those with blockage of the main heart arteries (triple vessel disease) to compare against.
* Participants in this pilot study will have additional tests used to diagnose CMD during their invasive angiography procedure. Participants will then have an MRI scan involving novel techniques and exercise MRI, where individuals exercise use a cycle or stepping machine during the MRI scan. Further analysis will also be undertaken of CT images acquired as part of the main study.
* These tests will be compared against invasive test results to see which show potential in being able to diagnose CMD.

DETAILED DESCRIPTION:
* Coronary artery disease (CAD) is the leading cause of morbidity and mortality in the United Kingdom. Approximately 40% of patients presenting with angina, however, have no evidence of significant obstructive CAD.
* About 60% of these patients have evidence of coronary microvascular disease (CMD), where there is dysfunction of the coronary microvessels leading to a mismatch between the blood supply to the myocardium and oxygen consumption. This may be due to a number of structural and functional changes including vascular remodelling, perivascular fibrosis, endothelial dysfunction and vascular smooth muscle dysfunction. Although previously thought of as a benign entity, recent studies suggest that CMD is associated with major adverse events.
* Symptoms caused by CMD and obstructive CAD cannot be distinguished sufficiently to guide diagnosis and management plans and conventional cardiac risk factors are poor discriminators of the two conditions, therefore clinicians are reliant on further investigations to diagnose CMD.
* Growing evidence supports invasive coronary physiological testing for this and methods to measure coronary vascular function during angiography have been developed. Once significant epicardial CAD has been excluded, CMD can be identified by impaired coronary flow reserve (CFR) and the index of microvascular resistance (IMR).
* Despite the ability of invasive testing to detect CMD, these methods come with attendant risks, as well as cost implications. Additionally, there is limited expertise and uptake amongst interventional cardiologists in intracoronary physiological assessment, limiting its widespread use. Hence, non-invasive surrogates are required to improve diagnosis and management of CMD. However, currently available non-invasive tests, including exercise ECG, stress echocardiography and nuclear imaging, lack the sensitivity and specificity to diagnose CMD.
* Microvascular volume analysed using novel imaging methods may provide the diagnostic accuracy required for the non-invasive identification of CMD. In CMD, patients may exhibit reduced microvascular volume, in contrast to epicardial disease where there is microvascular expansion and therefore these methods may be able to differentiate between the two disease processes. A number of methods have been proposed for assessment of microvascular volume using computed tomography (CT) and CMR. These methods include coronary luminal volume to myocardial mass (V/M) ratio using computational CT analysis, as well as CMR methods such as T1 mapping and Blood oxygen level-dependent CMR. Furthermore, compared to using pharmacological stress, exercise CMR could provide superior diagnostic ability to identify CMD, as it allows assessment during more 'physiological' stress.
* This study aims to provide pilot data on whether these novel CT and MRI and the use of physiological stress (exercise CMR) could identify CMD in patients presenting with angina. It aims to identify which of the proposed imaging methods could prove to be clinically useful for non-invasive identification of CMD, providing justification for a larger-scale diagnostic accuracy study.
* This is a prospective, single centre pilot study which will recruit individuals with angina referred for angiography who are participants in the research study 'CMR versus CT-FFR in CAD'.
* This pilot study will recruit both patients with suspected CMD and controls with multi-vessel CAD to compare against.
* Participants will be consented to have additional invasive testing at angiography for CMD. Those with confirmed CMD at angiography and all control participants will then have an MRI scan compromising of advanced MRI techniques for assessment of microvascular volume at rest and physiological stress (exercise). In addition, previously acquired CT images from the main research study will be transferred to Heartflow for computation of coronary blood volume.
* This will allow assessment of whether the novel imaging modalities proposed could be clinically useful for non-invasive identification of CMD and distinction from epicardial disease to inform larger future studies of these techniques.

ELIGIBILITY:
Inclusion Criteria:

* Current participant of the 'CMR versus CT-FFR in CAD' study
* Continue to meet the inclusion criteria for the main study:
* Patients aged ≥18 years
* Referred for invasive coronary angiography for investigation of chest pain
* Willing and able to give informed consent
* Willing and able (in the Investigators opinion) to comply with all study requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the study.
* Able to understand written English
* Able to perform exercise in the MRI scanner

Study arm:

* No evidence of obstructive or non-obstructive CAD on research CTCA
* Myocardial perfusion defect detected on adenosine stress CMR indicative of CMD

Control arm:

• Evidence of multivessel CAD on research CTCA

Exclusion Criteria:

* Meet the exclusion criteria for the main study:
* Recent acute coronary syndrome (< 6 months)
* Severe claustrophobia
* Absolute contraindications to CMR - those with MR conditional or safe devices will be included
* Second-/third-degree atrioventricular block
* Severe chronic obstructive pulmonary disease
* Moderate-severe asthma
* Estimated glomerular filtration rate <30 ml/min/1.73m2
* Women who are pregnant, breast-feeding or of child-bearing potential (premenopausal women)
* Contraindication to iodinated contrast
* Participants who have participated in a research study involving an investigational product in the past 12 weeks
* Patients unable to understand written English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected angina referred for invasive coronary angiography who are a current participants of the 'CMR versus CT-FFR in CAD' study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The ability of coronary luminal volume to myocardial mass (V/M) ratio measured using CT to identify the presence of CMD demonstrated by invasive coronary physiological assessment in patients with angina. | At time of imaging scan
The ability of T1 mapping at rest and exercise to identify the presence of CMD demonstrated by invasive coronary physiological assessment in patients with angina. | At time of imaging scan
The ability of Blood oxygen level-dependent CMR (BOLD-CMR) at rest and exercise at rest and exercise to identify the presence of CMD demonstrated by invasive coronary physiological assessment in patients with angina. | At time of imaging scan
The ability of CMR perfusion imaging at rest and exercise to identify the presence of CMD demonstrated by invasive coronary physiological assessment in patients with angina. | At time of imaging scan
The ability of myocardial blood volume as measured by CMR first-pass perfusion imaging at rest and during exercise to identify the presence of CMD demonstrated by invasive coronary physiological assessment in patients with angina. | At time of imaging scan

SECONDARY OUTCOMES:
T1 mapping at rest and adenosine-induced hyperaemia to identify the presence of CMD demonstrated by invasive coronary physiological assessment in patients with angina. | At time of imaging scan
CMR perfusion imaging at rest and adenosine-induced hyperaemia to identify the presence of CMD demonstrated by invasive coronary physiological assessment in patients with angina. | At time of imaging scan

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit Arnold, Principal Investigator — University of Leicester
Locations (1):
- Glenfield Hospital, University Hospitals of Leicester, Leicester, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided